CLINICAL TRIAL: NCT06307093
Title: International, Multicenter, Double-blind, Randomized, Comparative Study of the Pharmacokinetics, Safety and Efficacy of RPH-075 and Keytruda® in Patients With Malignant Neoplasms
Brief Title: Study Comparing the Pharmacokinetics, Safety, and Efficacy of RPH-075 and Keytruda® in Patients With Malignant Neoplasms
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Data Management 365 (Industry); Exacte Labs LLC (Industry); Federal State Budgetary Institution "NMIC of Hematology" of the Ministry of Health of the Russian Federation (Unknown); Federal State Budgetary Institution of the Central Research Institute of Epidemiology of Rospotrebnadzor (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL01860198
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Skin Melanoma; Squamous Non-small-cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: cancer; melanoma; carcinoma; lung cancer
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Neoplasms; Carcinoma; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPH-075 (Experimental): Pembrolizumab will be administered as an intravenous infusion every 3 weeks, at a fixed dose of 200 mg, for 30 minutes (it is permissible, but not desirable, to carry out an infusion in the range from 25 to 40 minutes).
  Premedication before administration of pembrolizumab is not mandatory.
  Interventions: Drug: RPH-075
- Keytruda® (Active Comparator): Pembrolizumab will be administered as an intravenous infusion every 3 weeks, at a fixed dose of 200 mg, for 30 minutes (it is permissible, but not desirable, to carry out an infusion in the range from 25 to 40 minutes).
  Premedication before administration of pembrolizumab is not mandatory.
  Interventions: Drug: Keytruda®

INTERVENTIONS:
Drug: RPH-075 — 100 mg/4 mL (25 mg/mL) concentrate for solution for infusions in a single-dose vial
  The required volume (8 ml) of the Drug concentrate solution should be withdrawn from the vials and transferred into an intravenous bag containing 0.9% Sodium Chloride Injection or 5% Dextrose Injection. (The final concentration of the diluted solution should be between 1 mg/mL to 10 mg/mL.)
  Other Names: pembrolizumab
  Arms: RPH-075
Drug: Keytruda® — 100 mg/4 mL (25 mg/mL) concentrate for solution for infusions in a single-dose vial
  The required volume (8 ml) of the Drug concentrate solution should be withdrawn from the vials and transferred into an intravenous bag containing 0.9% Sodium Chloride Injection or 5% Dextrose Injection. (The final concentration of the diluted solution should be between 1 mg/mL to 10 mg/mL.)
  Other Names: pembrolizumab
  Arms: Keytruda®

SUMMARY:
The goal of this double-blind, randomized study is to establish the equivalence of pharmacokinetic properties, as well as the comparability of safety, immunogenicity and pharmacodynamics of the drug RPH-075 (international nonproprietary name (INN) is pembrolizumab) in comparison with the drug Keytruda® (INN is pembrolizumab) after a single intravenous injection to patients with malignant neoplasms as a first or second line therapy in a monotherapy regimen.

The main main tasks are:

* To evaluate and compare the pharmacokinetic properties of RPH-075 and Keytruda® after a single intravenous administration of pembrolizumab to patients with malignant neoplasms;
* To evaluate the safety profile of the drug RPH-075 in comparison with the drug Keytruda® when used in patients with malignant neoplasms when used as a 1st or 2nd line therapy in a monotherapy regimen.

This study will also include a comparative assessment of immunogenicity, pharmacodynamic parameters and a pilot evaluation of RPH-075 efficacy.

DETAILED DESCRIPTION:
This study will include the following periods:

1. Screening period (before first administration of the test drug). Before being included in the study, patients will be provided with complete information about this clinical trial, its objectives, as well as the risks associated with participating in it, as set out in the patient information sheet.

   After the patient signs the Informed consent Form (IF), he will be examined as part of the screening period, at the end of which the researcher will decide whether or not the patient can be randomized into the study.
2. Main period (days: 1 - 168) Patients who meet the selection criteria will be randomized in a 1:1 ratio to one of the two study groups: RPH-075 and Keytruda®.

   Patients will receive pembrolizumab (RPH-075 or Keytruda®) in a monotherapy regimen, at a dose of 200 mg, intravenously, with a frequency of once every 3 weeks (3 weeks - 1 cycle). In case of significant adverse events (AEs), pembrolizumab therapy may be postponed for up to 12 weeks.

   Therapy within the Main Study period will continue until (whichever comes first):
   * 24 weeks (8 cycles);
   * disease progression (according to the Immune-Related Response Evaluation Criteria In Solid Tumors (iRECIST)/clinical progression);
   * the development of phenomena of intolerable toxicity.

   The assessment of tumor response to the therapy at this step will be carried out every 12 weeks.
3. Continued therapy period (days: 169 - 365) During the period of continued therapy, all patients will receive therapy with RPH-075, including those patients who received therapy with Keytruda® during the Main Study Period. Pembrolizumab will be administered intravenously, at a dose of 200 mg, with a frequency of once every 3 weeks. In case of significant AEs, pembrolizumab therapy may be postponed for up to 12 weeks.

   Therapy within the period of continued therapy will be carried out until (whichever comes first):
   * a period of up to 1 year;
   * before the disease progression (according to the criteria of iRECIST /clinical progression);
   * the development of phenomena of intolerable toxicity.

   The assessment of tumor response to the therapy at this step will be carried out every 12 weeks.
4. The period of further treatment (days: 366-730]) Participants in this period will be patients who, after 1 year of therapy, will have a stabilization of the disease or a tumor response to therapy. The decision to switch to this period wil be made by the researcher. If, according to the decision of the researcher, the patient will not be recommended to switch to this period, then the patient goes into the Follow-up Period.

   During the the period of further treatment patients will receive therapy with RPH-075 according to the same scheme as in the period of Continued therapy.

   Therapy within the Period will be carried out until (whichever comes first):
   * a total period of up to 2 years; all examinations will be carried out within the framework of routine clinical practice;
   * before the disease progression;
   * the development of phenomena of intolerable toxicity.

   All examinations necessary for the patient, including radiation diagnostics, and concomitant therapy during the Period will be carried out within the framework of routine clinical practice and through the healthcare system, with the exception of visits where therapy will be administered (every 3 weeks). Also, during these visits, data on the AEs and occurrence of events (progression) will be collected.
5. Follow-up period (FU)

For patients who will have completed their planned participation, namely:

* The period of further treatment,
* The period of continued therapy (those patients who will not be transferred during the pre-treatment Period),

one follow-up visit (FU-visit) will be scheduled 28 ± 3 days after the last administration.

For patients who will complete therapy ahead of schedule (within the Main period or the Period of continued therapy), due to the progression of the disease or the development of intolerant toxicity phenomena, FU visits will be conducted with a multiplicity of 1 every 12 weeks until the Day 365 of the study.

All examinations and concomitant therapy during the Follow-up Period will be provided through the health care system (as a part of routine clinical practice), with the exception of a radiation diagnostic visit conducting to assess the response (every 12 weeks).

The total expected duration of the study is approximately 3 years. The expected duration of participation of each subject is approximately 26 months (about 2 years).

ELIGIBILITY:
Inclusion Criteria:

1. A voluntarily signed and dated Informed Consent form (ICF) of the patient.
2. Histologically verified (there are documented results of relevant studies, in the absence of previous studies results, verification will be performed in the central laboratory) skin melanoma (patients with uveal melanoma or melanoma of the mucous membranes are not included in the study); squamous non-small cell lung cancer with Programmed death-ligand 1 (PD-L1) expression level ≥ 1% of tumor cells; head and neck squamous cell carcinoma with PD-L1 Tumor Proportion Score (TPS) expression level ≥ 50%.
3. The following patient populations:

   * with skin melanoma:

     * newly diagnosed, previously untreated, unresectable (stage III) or metastatic (stage IV) (the drug will be used as a 1st line therapy);
     * unresectable or metastatic, with progression during or after systemic antitumor therapy of the 1st line (the drug will be used as a therapy of the 2nd line);
     * with progression after previously performed neoadjuvant /adjuvant therapy, provided that the therapy was completed in a time exceeding 5 half-lives of the drug used, before randomization (the drug will be used as a 1-line therapy);
   * with squamous non-small-cell lung cancer:

     * newly identified unresectable (stage III) or metastatic (stage IV) with PD-L1 expression level ≥ 1%, with intolerance to 1st line chemotherapy (the drug will be used as 1st line therapy);
     * unresectable (stage III) or metastatic (stage IV) with PD-L1 expression level ≥ 1 %, with progression against the background of 1st line antitumor therapy (the drug will be used as a 2nd line therapy);
   * head and neck squamous cell carcinoma: • unresectable (stage III) or metastatic (stage IV) with PD-L1 TPS expression level ≥ 50% with progression during or after platinum-containing chemotherapy of the 1st line (the drug will be used as a therapy of the 2nd line).
4. The Eastern Cooperative Oncology Group (ECOG) score 0-2.
5. The presence of measurable control tumor foci (at least 1 focus), according to the Response evaluation criteria in solid tumors (RECIST) 1.1, confirmed by the conclusion of the Blinded Independent Central Response Assessment Committee.
6. Absence or resolution of toxic effects of previous therapy or negative consequences of surgical operations up to ≤ 2 grade according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0, with the exception of chronic / irreversible adverse events that do not affect the safety parameters of the studied therapy (for example, alopecia).
7. Life expectancy is at least 12 weeks from the date of randomization (according to the Researcher assessment).
8. Body weight: 50 to 100 kg.
9. Consent of female participants capable of childbirth, defined as all women with the physiological ability to conceive (with the exception of women with the final cessation of menstruation, which should be determined retrospectively after 12 months of natural amenorrhea, i.e. amenorrhea with an appropriate clinical status, for example, a suitable age), to use highly effective methods of contraception, starting with from the moment of signing the informed consent form and throughout the study (for at least 28 days after the last infusion of pembrolizumab) as well as the presence of a negative pregnancy test result (chorionic gonadotropin test). Consent of sexually active male participants in a clinical trial to use highly effective methods of contraception, starting from the moment of signing the informed consent form and throughout the study (for at least 28 days after the last infusion of pembrolizumab).

Exclusion Criteria:

1. Severe concomitant diseases, with life-threatening, acutely developing complications of the underlying disease (including massive pleural, pericardial or peritoneal effusion requiring aspiration, requiring intervention, pulmonary lymphangitis).
2. Metastases in the central nervous system, progressing or accompanied by clinical symptoms (for example, cerebral edema, spinal cord compression) or requiring the use of glucocorticosteroids (GCS) and/or anticonvulsants in doses specified in criterion No. 6; Patients with brain metastases can be included in the study if they receive adequate therapy (surgery or radiotherapy) and are stabilized by imaging studies for at least 4 weeks before the expected date of randomization into the study.
3. Concomitant diseases that are ongoing at the time of the screening examination and that increase the patient's risk of developing adverse events during the use of study therapy:

   * stable exertional angina of functional class III-IV, unstable angina, or a history of myocardial infarction suffered less than 1 month before the expected date of randomization into the study;
   * clinically significant rhythm disturbances (patients with asymptomatic atrial fibrillation can be included in the study provided the ventricular rhythm is controlled);
   * chronic heart failure of classes III-IV according to the New York Heart Association (NYHA) classification;
   * uncontrolled arterial hypertension (systolic blood pressure above 150 mmHg or diastolic blood pressure above 90 mmHg during antihypertensive therapy);
   * severe respiratory failure;
   * any other concomitant disease or condition that significantly increases the risk of developing adverse event (AE) during the study, in the opinion of the Investigator.
4. Systemic autoimmune diseases in the active phase (including, but not limited to: systemic lupus erythematosus (SLE), Crohn's disease, ulcerative colitis (UC), systemic scleroderma, inflammatory myopathy, mixed forms of connective tissue diseases, overlap syndrome, etc.), requiring systemic therapy for 2 years before expected date of randomization into the study.
5. Endocrine disorders that cannot be compensated for by regular hormone replacement therapy or other standard therapy at a constant dose for 28 days before the expected date of randomization into the study.
6. The need for therapy with GCS and any other drugs that have an immunosuppressive effect (at a dose equivalent to the daily use of prednisolone at a dose of >10 mg); the use of inhaled/topical drugs GCS is allowed; patients receiving Janus kinase (JAK) inhibitor therapy for coronavirus infection can be included in the study provided that JAK inhibitor therapy has been completed for at least 1.5 months. Before randomization, patients treated with anti-IL-6 drugs can be included in the study, provided that at least 5 half-lives of the anti-Interleukin 6 (IL-6) drug have passed before the expected date of randomization into the study.
7. Hematological disorders:

   * neutrophils < 1.5 x 10^9 /L,
   * platelets < 100 x 10^9 /L,
   * hemoglobin < 90 g/L.
8. Renal dysfunction:

   • creatinine > 1.5 × Upper limit of normal (ULN) or glomerular filtration rate < 45 ml/min.
9. Impaired liver function :

   * bilirubin ≥ 1.5 × ULN (except for patients with Gilbert's syndrome, whose total bilirubin values should not exceed 50 mmol/L),
   * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≥ 2.5 × ULN (5 × ULN for patients with liver metastases),
   * Alkaline phosphatase ≥ 5 × ULN
10. Conducting surgical treatment less than 28 days, radiation therapy less than 14 days before the expected date of randomization into the study.
11. Uveal melanoma or melanoma of the mucous membranes.
12. Possibility of radical removal of all metastatic foci.
13. Conducting 2 or more lines of systemic antitumor therapy for the underlying disease. (Prior therapy with targeted drugs (Serine/threonine-protein kinase B-raf (BRAF)/Mitogen-activated protein kinase (MEK) inhibitors, c-KIT (CD117) inhibitors) is allowed as 1st line therapy)
14. Previous therapy with pembrolizumab and other anti- Programmed cell death 1 (PD-1)/PD-L1/Programmed Cell Death 1 Ligand 2 (PD-L2) drugs.
15. The presence of another oncological pathology that is progressing or requires antitumor therapy (including hormonal) within 5 years before signing the ICF, with the exception of radically removed cervical carcinoma in situ, radically removed breast cancer in situ or radically removed basal cell/ squamous cell carcinoma of the skin.
16. Conditions that limit the patient's ability to comply with the requirements of the protocol (dementia, neurological or psychiatric disorders, drug and alcohol addiction, etc.).
17. Concurrent participation in other interventional clinical trials, participation in other clinical trials less than 30 days before signing the ICF (provided the patient has received at least one administration of experimental therapy), as well as previous participation in this clinical trial (provided the patient has received at least one administration of the drug RPH-075).
18. Acute infectious diseases or activation of chronic infectious diseases less than 28 days before the expected date of randomization into the study.
19. Active hepatitis B, hepatitis C, human immunodeficiency viruses (HIV) infection.
20. Therapy with live vaccines during the period 30 days before the expected date of randomization into the study. For patients receiving therapy with approved severe-acute-respiratory-syndrome-related coronavirus 2 (SARS-CoV2) vaccines, instructions for use and/or local requirements should be followed. The use of the Sputnik V vaccine is acceptable, provided that at least 7 days have passed from the moment of administration of the second component of the vaccine to the first administration of the study drug).
21. History of interstitial lung disease (non-infectious nature)/pneumonitis requiring the use of steroid therapy, current pneumonitis/Interstitial lung disease (ILD).
22. Impossibility of intravenous administration of the study drug.
23. Impossibility of intravenous contrast.
24. Hypersensitivity (grade 3 or more) to any of the components of the drug RPH-075/Keytruda®.
25. History of hypersensitivity to monoclonal antibody drugs.
26. Pregnancy or breastfeeding.
27. The presence of any other significant concomitant diseases or conditions that could, in the reasonable opinion of the study physician, adversely affect the patient's participation and well-being in the study and/or distort the evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Area under the curve "concentration-time" (AUC(0-504)) of pembrolizumab | pre-dose on Day 1 and 0, 2, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 336, 504 hours post-dose
  The area under the pharmacokinetic curve "concentration-time" of pembrolizumab after the first (single) administration, truncated to the second administration, i.e. the point 504 hours in both treatment groups.
Incidence of Adverse Reactions (ARs) | Days: 1 - 22
  Incidence of ARs in both treatment groups by system Organ Class or Preferred Term

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of pembrolizumab | pre-dose on Day 1 and 0, 2, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 336, 504 hours post-dose
  Pembrolizumab Cmax after the first administration in both treatment groups.
Maximum serum concentration of pembrolizumab at steady state (Сmax ss) | pre-dose on Day 106 (6th administration) and 0, 2, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 336, 504 hours post-dose
  Pembrolizumab C(max ss) after 6th administration in both treatment groups.
Minimal serum concentration of pembrolizumab at steady state (Сmin ss) | pre-dose on days: 43, 64, 85, 148
  Pembrolizumab C(min ss) after 6th administration in both treatment groups.
Area under the curve "concentration-time" of pembrolizumab at steady state (AUCtau ss) | pre-dose on Day 106 (6th administration) and 0, 2, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 336, 504 hours post-dose
  Area under the pharmacokinetic curve "concentration-time" of pembrolizumab at steady state (AUCtau ss) after 6th administration in both treatment groups.
Incidence of Treatment-Emergent Adverse Events (AEs) | Days: 1 - 168
  Incidence of treatment-emergent AEs in both treatment groups by system Organ Class or Preferred Term
Incidence of Immune-mediated adverse reactions (imARs) | Days: 1 - 168
  Incidence of imARs in both treatment groups by system Organ Class or Preferred Term
Incidence of Treatment-Emergent AEs with grade 3 or more | Days: 1 - 743 (up to 28 days after last pembrolizumab administration)
  Incidence of Treatment-Emergent AEs with grade 3 or more in both treatment groups by system Organ Class or Preferred Term
Incidence of Treatment-Emergent ARs with grade 3 or more | Days: 1 - 168
  Incidence of Treatment-Emergent ARs with grade 3 or more in both treatment groups by system Organ Class or Preferred Term
Incidence of imARs with grade 3 or more | Days: 1 - 168
  Incidence of imARs with grade 3 or more in both treatment groups by system Organ Class or Preferred Term
Incidence of serious adverse events (SAEs) | Days: 1 - 743 (up to 28 days after last pembrolizumab administration)
  Incidence of SAEs in both treatment groups by system Organ Class or Preferred Term
Incidence of serious adverse reactions (SARs) | Days: 1 - 168
  Incidence of SARs in both treatment groups by system Organ Class or Preferred Term
The proportion of patients (%) who required therapy discontinuation due to AR development | Days: 1 - 715
The proportion of patients (%) who developed binding antibodies and neutralizing antibodies to pembrolizumab | Days: 1, 22, 64, 106, 148

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (23):
- Russia (23):
  - State Budgetary Healthcare Institution of the city of Moscow "Moscow City Oncological Hospital No. 62 of the Department of Health of the City of Moscow", Istra, Moscow Oblast
  - "New Clinic" LLC, Pyatigorsk, Stavropol Territory
  - Regional State Budgetary Healthcare Institution "Altai Regional Oncological Dispensary", Barnaul, The Altai Republic
  - Autonomous Institution of the Chuvash Republic "Republican Clinical Oncological Dispensary" of the Ministry of Health of the Chuvash Republic, Cheboksary, The Chuvash Republic
  - State Autonomous Healthcare Institution Republican Clinical Oncological Dispensary of the Ministry of Health of the Republic of Bashkortostan, Ufa, The Republic of Bashkortostan
  - State Budgetary Healthcare Institution of the Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - Regional budgetary healthcare institution "Ivanovo Regional Oncological Dispensary", Ivanovo
  - State Budgetary healthcare Institution "Kuzbass Clinical Oncological Dispensary named after M.S. Rappoport", Kemerovo
  - State Budgetary Healthcare Institution of the city of Moscow "City Clinical Oncological Hospital No. 1 of the Department of Health of the City of Moscow", Moscow
  - State Budgetary Institution of Healthcare of the city of Moscow "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of the Department of Healthcare of the City of Moscow", Moscow
  - Federal State Budgetary Institution "N.N. Blokhin National Medical Research Center of Oncology" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Scientific Institution "Russian Scientific Center of Surgery named after Academician B.V. Petrovsky", Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - Medsi Group of Companies JSC, Moscow
  - "Research lab" LLC, Moscow
  - State Budgetary Healthcare Institution of the Perm Territory "Perm Regional Oncological Dispensary", Perm
  - State Budgetary Healthcare Institution Leningrad Regional Clinical Hospital, Saint Petersburg
  - Private healthcare institution "Clinical Hospital "Russian Railways-Medicine" of the city of St. Petersburg", Saint Petersburg
  - "Av Medical Group" LLC, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Clinical Oncological Dispensary", Saint Petersburg
  - Federal State Budgetary Institution "N.N. Petrov National Medical Research Center of Oncology" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - State Budgetary Healthcare Institution "Samara Regional Clinical Oncological Dispensary", Samara
  - The State Autonomous healthcare Institution of the Tyumen region "Multidisciplinary clinical Medical Center "Medical City", Tyumen